CLINICAL TRIAL: NCT03255278
Title: Evaluation of the Safety and Immunogenicity of the Recombinant Subunit Vaccine "GamTBvac" Against the Tuberculosis. Comparative Placebo-controlled Study With a Two-fold Increase of the Vaccine Dose in Healthy Volunteers Aged 18-49 Years.
Brief Title: Evaluation of the Safety and Immunogenicity of the Recombinant Subunit Vaccine "GamTBvac" Against the Tuberculosis.
Acronym: GamTBvac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: GamTBvac Ph1
Record Dates: First submitted 2017-06-29; First posted 2017-08-21 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Recombinant vaccine; Mycobacterium tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: The clinical trial study of the "GamTBvac" vaccine against the tuberculosis is a comparative placebo-controlled study with a two-fold increase of an applied dose among healthy volonteers aged 18-49 years.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Safety and portable study group (Experimental): 12 persons who have got a single decreased dose (0.25 of the planned dose for regular administration) of the GamTBvac recombinant subunit vaccine.
  The intervention for the Arm: single GamTBvac vaccination (0.25 dose).
  Interventions: Biological: Single GamTBvac vaccination (0.25 dose)
- Placebo safety study group (Placebo Comparator): 12 persons who have got a single dose of placebo (0.5 ml). The intervention for the Arm: Placebo administration (0.5 ml)
  Interventions: Biological: Placebo administration
- Immunogenicity study group #1 (Experimental): 12 persons who will get a double sequential administration of the decreased dose (0.25 of the planned dose for regular applying) of the GamTBvac recombinant subunit vaccine.
  The intervention for the Arm: double GamTBvac vaccination (0.25 dose).
  Interventions: Biological: Double GamTBvac vaccination (0.25 dose)
- Immunogenicity study group #2 (Experimental): 12 persons who will get a double sequential administration of the mean dose (0.5 of the planned dose for regular applying) of the GamTBvac recombinant subunit vaccine.
  The intervention for the Arm: double GamTBvac vaccination (0.5 dose).
  Interventions: Biological: Double GamTBvac vaccination (0.5 dose)
- Immunogenicity study group #3 (Experimental): 12 persons who will get a double sequential administration of the maximum (regular) dose of the GamTBvac recombinant subunit vaccine.
  The intervention for the Arm: double GamTBvac vaccination (1.0 dose).
  Interventions: Biological: Double GamTBvac vaccination (1.0 dose)

INTERVENTIONS:
Biological: Single GamTBvac vaccination (0.25 dose) — Single administration of the decreased dose of vaccine (0.25 of regular dose) to evaluate the safety.
  Arms: Safety and portable study group
Biological: Placebo administration — Single administration of the placebo (0.5 ml) to a placebo safety study group (Arm 2).
  Arms: Placebo safety study group
Biological: Double GamTBvac vaccination (0.25 dose) — Double sequential administration of the decreased dose of vaccine (0.25 of regular dose) to evaluate the immunogenicity.
  Arms: Immunogenicity study group #1
Biological: Double GamTBvac vaccination (0.5 dose) — Double sequential administration of the mean dose of vaccine (0.5 of regular dose) to evaluate the immunogenicity.
  Arms: Immunogenicity study group #2
Biological: Double GamTBvac vaccination (1.0 dose) — Double sequential administration of the regular dose of vaccine to evaluate the immunogenicity.
  Arms: Immunogenicity study group #3

SUMMARY:
The study is aimed to evaluate the safety and immunogenicity of the medicinal product "GamTBvac" - a recombinant subunit vaccine against the tuberculosis. The study is designed as a comparative placebo-controlled study with a two-fold increase of an applied dose among healthy volunteers aged 18-49 years.

DETAILED DESCRIPTION:
The clinical trial study of the "GamTBvac" vaccine against the tuberculosis is a comparative placebo-controlled study with a two-fold increase of an applied dose among healthy volunteers aged 18-49 years. The product "GamTBvac" is a lyophilized substance consisted of the purified recombinant subunit antigens of Mycobacterium tuberculosis, that is applied for the preparing of the solution for a subcutaneous administration. Currently the study is at the first phase.

The aims of the study are: a) to confirm the safety of the product in the healthy volunteers; b) to select the optimal administration dose; c) to evaluate of the immunogenicity of the vaccine; d) to investigate the immune cell memory as a response to the vaccination.

The total number of the volunteers in the study is 60:

1. at the first stage to estimate the safety and portable of the vaccine, two groups of volunteers each includes 12 persons got the single decreased dose (0.25 of the planned dose for regular administration) of the vaccine (the first group, 12 persons), and the 0.5 ml of the placebo (the second group, 12 persons);
2. at the second stage to select the optimal dose and the scheme of the vaccine administration, additionally three groups, each consist of 12 persons of volunteers will be recruited. The first group will get double vaccination of a decreased dose (0.25 of the regular dose), the second group will get the double vaccination of a mean dose (0.5 of the regular dose), and the third one will get the double vaccination of the maximum (1.0 regular) dose.

The inclusion criteria for the volunteers of the study are: healthy males either females aged 18-49 years who have previously got the BCG vaccine. The exclusion criterion is the presence of the latent tuberculosis in the patient that is confirmed during the preliminary laboratory screening.

ELIGIBILITY:
Inclusion Criteria:

* lack of the latent tuberculosis, laboratory confirmed
* BCG vaccination in the past
* signed informed consent

Exclusion Criteria:

* presence of the latent tuberculosis, laboratory confirmed

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
The number and severity of adverse effects | 140 Days
  Safety control: an active periodical examination of the health status of volunteers, including vital indicators, instrumental tests (ECG), laboratory blood and urine analysis (general and biochemistry). The presence, nature and severity of local and systemic reactions in different groups of volunteers, depending on the dose of vaccination, will be taken into account.

SECONDARY OUTCOMES:
immunogenicity control | 140 Days
  Qualitative ELISA test for specific IgG antibodies, study of the stimulated T-cell

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tkachuk AP, Gushchin VA, Potapov VD, Demidenko AV, Lunin VG, Gintsburg AL. Multi-subunit BCG booster vaccine GamTBvac: Assessment of immunogenicity and protective efficacy in murine and guinea pig TB models. PLoS One. 2017 Apr 28;12(4):e0176784. doi: 10.1371/journal.pone.0176784. eCollection 2017. PMID 28453555
- See also: Tkachuk AP, Gushchin VA, Potapov VD, Demidenko AV, Lunin VG, Gintsburg AL. Multi-subunit BCG booster vaccine GamTBvac: Assessment of immunogenicity and protective efficacy in murine and guinea pig TB models. PLoS One. 2017 Apr 28 — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0176784